CLINICAL TRIAL: NCT05821127
Title: The Effect of Neurodynamic Exercises and Education Program Applied With Virtual Reality Assisted Telerehabilitation Method in Conservative Treatment of Carpal Tunnel Syndrome: A Single-Blind Randomized Controlled Trial
Brief Title: Effect of Neurodynamic Exercises and Education Program Applied With Virtual Reality Assisted Telerehabilitation Method in Conservative Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Baran Sezgin, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Istanbul University, Turkey
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Carpal Tunnel Syndrome; Peripheral Neuropathy; Median Nerve Entrapment
Keywords: Carpal Tunnel Syndrome; Virtual Reality; Telerehabilitation; Exercise; Education; Ergonomics
MeSH Terms: conditions — Carpal Tunnel Syndrome; Peripheral Nervous System Diseases; Median Neuropathy; Motor Activity | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: A random number table containing numbers from 1 to 60 was created for 2 groups through the computer program. Participants were numbered in order of application. Participants were assigned to groups to which their numbers belonged in the table of random numbers.
Who Masked: Outcomes Assessor
Masking Description: It was noted to which group the patient was allocated by referring to the list of random numbers created by a computer program by a researcher participating in the study. The treatment process for the intervention group and the control group was managed by the same researcher. Outcome evaluations before treatment and after 8 weeks of treatment follow-up were made by a second researcher who was blind to group distribution. The list of random numbers was hidden from the researcher making the evaluations, ensuring that the participants did not know which group they belonged to. Analysis of the data was done by a third researcher. The intervention group was coded as 'group 1' and the control group was coded as 'group 2'. With this method, it was ensured that the researcher performing the analysis did not know which group the patients belonged to. With this randomization and blinding process, the impartiality of the researchers was ensured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Assisted Neurodynamic Exercises and Patient Education with Telerehabilitation Method (Experimental): Patient education was provided in 3 sessions via telerehabilitation method, and exercises were provided with virtual reality support. It was requested that the exercises be done in 6 sets (30 repetitions) every day. Participants were given a splint, exercise brochure, and exercise diary for use at night.
  Interventions: Behavioral: Virtual Reality Assisted Neurodynamic Exercises and Patient Education with Telerehabilitation Method
- Neurodynamic Exercises and Patient Education with Traditional Method (Active Comparator): Participants were given a single session of face-to-face training on the same topics, and were given a splint, exercise brochure and exercise diary to be used at night.
  Interventions: Behavioral: Neurodynamic Exercises and Patient Education with Traditional Method

INTERVENTIONS:
Behavioral: Virtual Reality Assisted Neurodynamic Exercises and Patient Education with Telerehabilitation Method — A brochure showing the execution of median nerve and tendon gliding exercises and a wrist brace for night use will be provided. In addition, 2 sessions of patient education will be provided with videoconference calls, and with the mobile application to be installed on the phones of the patients as non-immersive virtual reality support, it will be possible to practice median nerve and tendon gliding exercises in the form of 5 repetitions and 6 sets every day with video support for 16 weeks. In this application, the user will use the front camera of phone as a sensor to detect hand movements. A screen on which exercises will be played at the top of the screen and a virtual image of the user's hand in the lower half of the screen will be displayed in the field of view of the camera. Each exercise position will take 5 seconds. Patient education will include neuroscience, etiology, pathophysiology and treatment options of carpal tunnel syndrome, ergonomics and posture education.
  Arms: Virtual Reality Assisted Neurodynamic Exercises and Patient Education with Telerehabilitation Method
Behavioral: Neurodynamic Exercises and Patient Education with Traditional Method — A brochure showing the execution of median nerve and tendon gliding exercises and a wrist brace for night use will be provided. Patients will be asked to do the exercises in the form of 5 repetitions and 6 sets every day and to wear the night splint every night for 16 weeks. Each exercise position will take 5 seconds. A brief verbal education will be given to the patients under the same topics as the intervention group, as in the outpatient clinic.
  Arms: Neurodynamic Exercises and Patient Education with Traditional Method

SUMMARY:
The aim in this prospective, randomized and controlled, single-blind study; In the conservative treatment of patients diagnosed with carpal tunnel syndrome, to investigate the effects of neurodynamic exercises that applied with nonimmersive virtual reality technology and patient education program presented by the telerehabilitation method on pain-numbness, functional status and quality of life, to compare the effects of neurodynamic exercises that applied with traditional methods and standard education given to patients in outpatient clinic conditions on the same parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Being diagnosed with CTS clinically and electrophysiologically

Exclusion Criteria:

* <18 years or >65 years
* Distal motor latency > 6.0 msn.
* Thenar atrophy
* Surgery history for CTS
* Steroid injection for CTS
* Physical treatment for CTS in the last 6 months
* Cervical radiculopathy
* Tenosynovitis
* Peripheral polyneuropathy
* Another compressive neuropathy in the ipsilateral upper extremity
* History of trauma/fracture to the hand-wrist region
* Pregnancy
* Metabolic disease
* Rheumatic/autoimmune disease
* Kidney failure
* Lack of internet access
* Not having the equipment to make video calls at home

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Syndrome Questionnaire (BCTSQ) | baseline, eight week of intervention, sixteen week of intervention
  BCTSQ assesses the severity of symptoms and functional status in patients with carpal tunnel syndrome. The symptom severity scale assesses the symptoms with respect to severity, frequency, time and type. The scale consists of 11 questions with multiple-choice responses, scored from 1 point (mildest) to 5 points (most severe). The overall symptom severity score is calculated as the mean of the scores for the eleven individual items. The functional status scale assesses the affect of the carpal tunnel syndrome on daily living. The scale consists of 8 questions with multiple choice responses, scored from 1 point (no difficulty with the activity) to 5 points (can not perform the activity at all). The overall score for functional status was calculated as the mean of all eight. Thus, a higher symptom severity or functional status score indicates worse symptoms or dysfunction.
Change in Visual Pain Scale (VAS) | baseline, eight week of intervention, sixteen week of intervention
  The VAS is a single-item measure, that is, an instrument measuring the whole construct at once. VAS most commonly consists of a 100mm horizontal line anchored with two opposite labels; patients mark a score on the scale using a vertical line. Using this scale, patients will be asked to rate the severity of pain and numbness they feel during the night and in daytime at rest, and with activity between 0 and 100 points.

SECONDARY OUTCOMES:
Change in Brief International Classification of Functioning (ICF) Core Set for Hand Conditions Questionnaire | baseline, eight week of intervention, sixteen week of intervention
  The disorders caused by carpal tunnel syndrome in the patient's daily activities will be evaluated by using the 'ICF activities and participation codes' section of the 'Brief ICF Core Set for Hand Conditions'.
Change in Short Form-36 (SF-36) Questionnaire | baseline, eight week of intervention, sixteen week of intervention
  The SF-36 is a 36 item questionnaire that measures eight multi-item dimensions of health: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy/vitality, pain and general health perception. For each dimension item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state).
Change in Semmes Weinstein Monofilament Test (SWMT) | baseline, eight week of intervention, sixteen week of intervention
  Using 20 pieces of SWMT, sensitive touch threshold sensitivity of each hand will be tested. The examiner and the subject will seated opposite each other. Both arms of the subject will arranged on a table in supination, with palm upwards. The patient will be instructed to close their eyes. The monofilaments will be touched fingertips of first three fingers on the radial side of both hands, with enough force to bend the monofilament for 1.5 seconds. The thinnest monofilament numbers that the patient feels being touched will be recorded. The thinnest monofilament number among the three measurements will be noted as a result. Absence of sensation at a threshold of 2.83 in any of the three fingers tested indicates loss of sensation.
Change in Two Point Discrimination Test (TPDT) | baseline, eight week of intervention, sixteen week of intervention
  Two point discrimination sense will be evaluated statically and dynamically using an esthesiometer. The examiner and the subject will seated opposite each other. Both arms of the subject will arranged on a table in supination, with palm upwards. The patient will be instructed to close their eyes. The contact time of the discriminator with the fingertip ranged from 3 to 5 seconds. The evaluation will be started by touching a single point on the first three fingertips on the radial side of both hands. Each three fingers will be evaluated separately and the distance between the two touched points will be increased by 1mm in each measurement. The smallest values will be taken in millimeters which the patient feels the two points as two separate points on the tested hand will be noted and the the average value written as the result.
Change in Hand Grip Force | baseline, eight week of intervention, sixteen week of intervention
  The squeeze force will be measured while the patients are sitting, with the elbow in 90 degrees flexion and they will be asked to make a maximally voluntary grip. Measurements will be made three times in a row on both hands and the average of the three measurements will be noted as a result in kilogram (kg).
Change in Thumb and Forefinger Pinch Force | baseline, eight week of intervention, sixteen week of intervention
  The pinch force with thumb and forefinger will be measured while the patients are sitting, with the elbow in 90 degrees flexion and they will be asked to make a maximally voluntary grip.The pinch force will be measured as kg with a pinch dynamometer, and the average of the three measurements will be noted as a result.
Change in Manuel Muscle Testing of M. Abductor Pollicis Brevis | baseline, eight week of intervention, sixteen week of intervention
  Manual muscle testing will be evaluated in 5 grades. No visible or palpable muscle contraction 0, visible or palpable muscle contraction without motion grade 1, muscle contraction that creates movement at full of range of motion when gravity is eliminated grade 2, muscle contraction that creates movement at full of range of motion against gravity grade 3, muscle contraction that creates movement at full of range of motion against gravity and moderate resistance grade 4, muscle contraction that creates movement through the entire range of motion of the joint against gravity and full resistance will be considered as the grade 5.
Change in Vibration Sensation | baseline, eight week of intervention, sixteen week of intervention
  Vibration sense was tested with tuning fork. The normal vibration sensory threshold for the upper extremity was accepted as 20 seconds. The examiner and the subject will seated opposite each other. Both arms of the subject will arranged on a table in supination, with palm upwards. The patient will be instructed to close their eyes. Vibrating tuning fork will be placed on the palmar aspect of the distal phalanx of first three fingers on the radial side of both hands, The patient was asked to say 'done' when the vibration in his hand was over. The average of three measurements will be noted as a result in seconds.
Change in Nerve Conduction Study (NCS) | baseline, eight week of intervention, sixteen week of intervention
  Median motor distal latency and conduction velocity and second finger recorded median sensory distal latency and conduction velocity will be measured antidromically in all individuals. In addition to routine conduction examinations, fourth finger recorded median-ulnar peak latency comparison examinations will also be made.

CONTACTS AND LOCATIONS:
Overall Officials: Baran Sezgin, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No